CLINICAL TRIAL: NCT03231930
Title: Rapid Point-of-care Testing for Hepatitis C in Community Clinics (RAPID-EC) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/16/Alfred/165
Record Dates: First submitted 2017-06-25; First posted 2017-07-27 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
Keywords: Diagnosis; Point of Care Diagnostics; Hepatitis
MeSH Terms: conditions — Hepatitis C; Disease; Hepatitis

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention, which is rapid point of care testing for hepatitis C antibodies using the OraQuick test with oral fluid , followed by point of care testing for the detection of hepatitis C virus RNA using the Cepheid Xpert HCV RNA viral load test on the GeneXpert system. Participants who are found to have current HCV infection will be worked up for treatment at ths clinic and referred to appropriate practitioners for HCV treatment. All results will be confirmed with standard laboratory testing as these devices are not yet approved for diagnostic use in Australia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention group (Experimental): Rapid point of care testing will be done using the OraQuick HCV Ab test and the Xpert HCV RNA viral load test. All participants will undergo rapid point of care testing for hepatitis C antibodies using the OraQuick test with oral fluid, followed by point of care testing for the detection of hepatitis C virus RNA using the Cepheid Xpert HCV viral load test on the GeneXpert system. Participants who are found to have current HCV infection will be worked up for treatment at the clinic and referred to appropriate practitioners for HCV treatment. As these tests are not yet licensed for diagnostic use in Australia, confirmatory testing using standard laboratory tests will be performed for all participants.
  Interventions: Device: OraQuick HCV Ab test; Device: Xpert HCV viral load test

INTERVENTIONS:
Device: OraQuick HCV Ab test — The OraQuick HCV point of care test involves the collection of oral fluid and provides an accurate result in approximately 20 minutes. The test involves a clinic nurse or community health worker providing pre-test counselling, then providing an oral swab to study participants, then reading the result and counselling the participant about their HCV antibody test result.
Device: Xpert HCV viral load test — The Cepheid Xpert HCV RNA test (Xpert® HCV Viral Load test) is a reverse transcriptase polymerase-based chain reaction amplification technology (RT-PCR) and provides an accurate HCV RNA load within 2 hours (105 minutes), using a serum sample.
  This test will be performed for participants who have a positive OraQuick HCV antibody result.

SUMMARY:
The Rapid-EC pilot study will determine feasibility of providing rapid point-of-care (POC) testing for HCV in community clinics, and whether the availability of POC testing increases uptake of testing, engagement in care and completion of treatment among people who inject drugs.

The POC tests being utilised in this study are the OraQuick mouth swab test for the presence of HCV antibodies, and the Xpert HCV RNA viral load test using serum.

DETAILED DESCRIPTION:
The introduction of direct-acting antiviral (DAA) therapies has meant the elimination of hepatitis C (HCV) as a public health issue in Australia is a very real possibility. The challenge that remains is to ensure that all people living with HCV can access testing to become aware of their status, and then get treated and cured. Given that people who inject drugs (PWID) account for the vast majority of new HCV infections in Australia, this group will be key to elimination efforts. Innovative approaches are needed to overcome the barriers to accessing health services that are faced by PWID.

The Rapid-EC pilot study will determine feasibility of providing rapid point-of-care (POC) testing for HCV in community clinics, and whether the availability of POC testing increases uptake of testing, engagement in care and completion of treatment among PWID.

The Rapid-EC pilot study will be delivered by a multi-disciplinary team in three community clinics in Melbourne, Australia. After providing informed consent and receiving pre-test counselling, participants will undergo an OraQuick mouth swab test for the presence of HCV antibodies, which indicates whether a person has ever been exposed to HCV. This result is available in 20 minutes. If this test is positive they will then be offered a test for the presence of virus in the blood, known as a PCR or RNA test. The Xpert HCV RNA POC test uses a 5ml sample of blood from the vein and is run on the GeneXpert machine, which will be on-site at each clinic. This machine provides results in 105 minutes, allowing participants to receive a HCV diagnosis on the day of testing.

Both the OraQuick HCV Ab test and the Xpert HCV RNA test are highly accurate tests; however they are currently awaiting approval for diagnostic use in Australia. As such, standard-of-care testing will be performed for all participants to confirm the result and inform clinical care. Participants who have a positive HCV Ab result will have a follow-up visit with the study nurse where they will review all test results. Those who are found to have a current HCV infection (positive RNA result) will have an assessment of liver health and, where appropriate, commence HCV treatment from the clinic. Participants will be reimbursed for the time taken to complete the study.

To evaluate the impact of the study participants will be asked to complete two questionnaires: 1) at the beginning of the study to record demographics, risk behaviours, and previous experience of HCV testing; and 2) after completing the POC tests to provide feedback on their experience and preferences for testing. These responses, as well as clinical information collected by staff, will be de-identified. Data linkage with Medicare and Pharmaceutical Benefits Scheme data will be used to determine if the participant followed up with their healthcare provider and collected a prescription for HCV treatment.

This study will provide valuable insights into the feasibility and effects of offering POC testing for HCV, particularly the effect on uptake of testing and treatment. The results will inform a larger trial, with greater numbers of participants and sites, and the introduction of finger prick testing for HCV RNA, which is likely to become available for research use in towards the end of 2017.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Attendance for any reason at either the primary health care services participating in the study
* Not currently engaged in care for treatment of hepatitis C infection, and not received a diagnosis of hepatitis C infection (with positive HCV RNA) in the preceding 3 months;

Exclusion Criteria:

* Pregnancy or breastfeeding at time of HCV antiviral treatment;
* Evidence of any condition, therapy, laboratory abnormality or other circumstance (current or prior) that may confound the study's results, or interfere with participation for the full duration of the study, such that it is not in the best interest of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Number of participants at high risk for HCV infection who receive a HCV rapid point-of-care antibody test | 6 months after commencing recruitment.
  The investigators will measure the total number of participants who undergo the OraQuick test for HCV antibodies. This will be recorded by site staff.

SECONDARY OUTCOMES:
Number of participants with a positive HCV antibody test who receive a rapid point-of-care RNA test | 6 months after commencing recruitment.
  The investigators will measure the total number of participants who undergo the Xpert HCV viral load test for HCV RNA. This will be recorded by site staff.
Number of participants with a positive HCV RNA test who attend their appointment with the doctor for treatment | 6 months after commencing recruitment.
  The investigators will measure how many participants attend a follow-up appointment with their doctor to discuss treatment. This will be recorded by site staff.
Number of participants who obtain DAA therapy (ie medication is picked up from pharmacy) | Six months post completion of recruitment
  The investigators will measure the number of participants who collect medication for treatment by accessing data from the Pharmaceutical Benefits Scheme, with participant consent.
Number of participants who achieve sustained virological response at 12 weeks post treatment (SVR12) | Six months post completion of recruitment
  This will be measured using standard of care blood tests for HCV RNA at 12 weeks post completion of treatment, with results reviewed and recorded by site staff.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hellard, MBBS,PhD, Principal Investigator — Burnet Institute
Locations (3):
- Australia (3):
  - Innerspace, Collingwood, Victoria
  - Health Works, Footscray, Victoria
  - North Richmond Community Health, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Williams B, Howell J, Doyle J, Thompson AJ, Draper B, Layton C, Latham N, Bramwell F, Membrey D, Mcpherson M, Roney J, Stoove M, Hellard ME, Pedrana A. Point-of-care hepatitis C testing from needle and syringe programs: An Australian feasibility study. Int J Drug Policy. 2019 Oct;72:91-98. doi: 10.1016/j.drugpo.2019.05.012. Epub 2019 May 22. PMID 31129023
- [Result] Latham NH, Pedrana A, Doyle JS, Howell J, Williams B, Higgs P, Thompson AJ, Hellard ME. Community-based, point-of-care hepatitis C testing: perspectives and preferences of people who inject drugs. J Viral Hepat. 2019 Jul;26(7):919-922. doi: 10.1111/jvh.13087. Epub 2019 Apr 1. PMID 30801881